CLINICAL TRIAL: NCT05861830
Title: An Exploratory Study on Predicting the Efficacy of Dalpiciclib in Combination With Endocrine Therapy for HR-Positive and HER2-Negative Recurrent/Metastatic Breast Cancer Patients After CDK4/6 Inhibitor Treatment Failure Using 18F-FES PET/CT
Brief Title: Dalpiciclib With Endocrine Therapy for Advanced Breast Cancer After CDK4/6 Inhibitor Failure (DAWNA-FES)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUMCH-FES-BC-2
Record Dates: First submitted 2023-05-07; First posted 2023-05-17 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): The combination of Dalpiciclib with physician-selected endocrine therapy
  Interventions: Drug: The combination of Dalpiciclib with physician-selected endocrine therapy
- Arm B (Active Comparator): Chemotherapy selected by the physician
  Interventions: Drug: Chemotherapy selected by the physician

INTERVENTIONS:
Drug: The combination of Dalpiciclib with physician-selected endocrine therapy — * Dalpiciclib: 150 mg, orally, once daily, on days 1-21, every 28 days (3 weeks on, 1 week off)
  * Letrozole: 2.5 mg, orally, once daily (continuous), every 28 days OR Anastrozole: 1.0 mg, orally, once daily (continuous), every 28 days OR Exemestane: 25 mg, orally, once daily (continuous), every 28 days OR Fulvestrant: 500 mg, intramuscular injection on day 1/15 of the first cycle, then on day 1 of each subsequent cycle, every 28 days OR Tamoxifen: 10-20 mg, orally, twice daily (continuous), every 28 days
  * Pre/perimenopausal women also require ovarian function suppression (OFS), which can be achieved through bilateral oophorectomy or the use of gonadotropin-releasing hormone (GnRH) analog drugs
  Arms: Arm A
Drug: Chemotherapy selected by the physician — The chemotherapy regimen is chosen by the clinical physician and may include, but is not limited to, the following options: the combination of paclitaxel and capecitabine, the combination of paclitaxel and carboplatin, single-agent capecitabine, single-agent platinum drugs, and the combination of gemcitabine and platinum-based chemotherapy. Each treatment cycle consists of a 21-day duration.
  Arms: Arm B

SUMMARY:
CDK4/6 inhibitors are currently the standard treatment for female breast cancer patients with HR+ tumors. However, there is no established standard treatment for patients who experience treatment failure with CDK4/6 inhibitors. The MAINTAIN study has shown clinical benefits by switching to Ribociclib and changing endocrine therapy after progression on CDK4/6 inhibitors. We hypothesize that combining Dalpiciclib with physician-selected endocrine therapy, following treatment failure with CDK4/6 inhibitors, would similarly lead to improved patient survival. In this study, 18F-FES PET/CT will be employed as a non-invasive alternative to biopsy techniques for evaluating the expression of ER in various systemic lesions of the patients.

DETAILED DESCRIPTION:
With the emergence of targeted therapies, the treatment landscape for patients with hormone receptor-positive (HR+) and HER2-negative (HER2-) metastatic breast cancer (MBC) is continuously evolving. The combination of cyclin-dependent kinases 4 and 6 inhibitors (CDK4/6i) with endocrine therapy has become the standard treatment approach for first-line therapy or treatment after progression on endocrine therapy. Multiple large randomized studies have demonstrated that the combination of CDK4/6i and endocrine therapy significantly improves progression-free survival (PFS) in HR+/HER2- MBC patients. Updated analyses have also shown a significant improvement in overall survival (OS) with the combination of endocrine therapy and either Palbociclib or Ribociclib. Currently, regulatory agencies have approved four CDK4/6 inhibitors, namely Palbociclib, Abemaciclib, Ribociclib, and Dalpiciclib, for the treatment of HR+/HER2- breast cancer. All four CDK4/6 inhibitors are approved for use in combination with endocrine therapy for advanced HR+/HER2- breast cancer. Abemaciclib has also been approved for use as adjuvant therapy in early-stage breast cancer with HR+/HER2- subtype and high-risk recurrent factors, as well as for the treatment of advanced breast cancer.

CDK4/6 inhibitors are currently the standard treatment for female breast cancer patients with HR+ tumors. However, there is no established standard treatment for patients who experience treatment failure with CDK4/6 inhibitors. Despite the extensive clinical experience with these drugs, our understanding of the long-term effects of CDK4/6 blockade in patients previously treated with CDK4/6 inhibitors is limited. The MAINTAIN study has shown clinical benefits by switching to Ribociclib and changing endocrine therapy after progression on CDK4/6 inhibitors. We hypothesize that combining Dalpiciclib with physician-selected endocrine therapy, following treatment failure with CDK4/6 inhibitors, would similarly lead to improved patient survival.

18F-fluorodeoxyglucose (FDG) PET imaging is widely utilized in the field of oncology to detect increased glucose metabolism activity. In the case of breast cancer, 18F-FDG PET/CT imaging is predominantly recommended for patients with unclear staging, advanced disease, or metastasis, when conventional imaging methods are inconclusive. On the other hand, 18F-fluoroestradiol (FES) is an endogenous estrogen analogue that specifically binds to estrogen receptors (ERs). Through PET imaging, FES enables dynamic, quantitative, and non-invasive assessment of ER expression levels and distribution within the patient's body. When combined with 18F-FDG PET or other imaging modalities, 18F-FES PET imaging can evaluate the heterogeneity of ER expression and has the potential to identify ER loss or dysfunction. It has been observed that 18F-FES PET exhibits good correlation with traditional immunohistochemistry for assessing ER expression. Moreover, published human studies have not reported any toxicity or adverse reactions associated with 18F-FES usage. In this study, 18F-FES PET/CT will be employed as a non-invasive alternative to biopsy techniques for evaluating the expression of ER in various systemic lesions of the patients.

ELIGIBILITY:
Inclusion Criteria:

* The recent pathology results showed HR-positive and HER2-negative.
* 18F-FES-PET/CT showed at least one ER-positive lesion.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score: 0-2 points.
* Expected survival time ≥ 3 months.
* Previous antitumor therapy: (1) (neo)adjuvant treatment with Palbociclib or Abemaciclib or Ribociclib or relapse after adjuvant treatment with Palbociclib or Abemaciclib or Ribociclib; (2) receiving Palbociclib or Abemaciclib or Ribociclib-based treatment in the context of metastatic breast cancer or disease progression after treatment; (3) previously received ≤1 line of chemotherapy for recurrent or metastatic breast cancer; (4) previously received ≤3 lines of endocrine therapy for recurrent or metastatic breast cancer.
* Willing to undergo 18F-FDG PET/CT standard imaging.
* At least one measurable lesion outside the skull according to RECIST V1.1.
* The function of important organs meets the requirements.
* The subjects have recovered from any adverse event related to previous tumor treatment (≤ Grade 1) before the first administration of the investigational drug.

Exclusion Criteria:

* 18F-FES-PET/CT shows that all lesions are ER-negative.
* Previously received treatment with Dalpiciclib.
* MRI or lumbar puncture confirms leptomeningeal metastasis.
* Imaging confirms central nervous system metastasis.
* Participants with visceral crisis, rapid disease progression, and patients not suitable for endocrine therapy.
* Participants with ascites, baseline pleural effusion with clinical symptoms, and pericardial effusion requiring drainage within the first 4 weeks of treatment.
* Unable to swallow, intestinal obstruction, or other factors that affect drug administration and absorption.
* Participants diagnosed with any other malignancy within the past 5 years, excluding non-melanoma skin cancer treated with curative intent. Basal cell or squamous cell skin cancer, or cervical intraepithelial neoplasia and papillary thyroid cancer.
* Participants who have undergone major surgery or suffered a major injury within 4 weeks before starting treatment, or are expected to undergo major surgical treatment.
* Known history of allergy to the components of this treatment regimen.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed PFS | Up to approximately 24 months
  The time from the initiation of treatment to the first radiographic assessment of disease progression (PD) or any event leading to death

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective Response Rate
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate
Overall Survival (OS) | Up to approximately 24 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Sun, M.D., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China